CLINICAL TRIAL: NCT04142307
Title: Biofeedback in Idiopathic Infantile Nystagmus Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monica Daibert Nido (Other)
Responsible Party: Sponsor-Investigator, Monica Daibert Nido, Assistant Professor, University of Toronto
Organization: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Biofeedback Low Vision
Record Dates: First submitted 2019-10-22; First posted 2019-10-29 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Low Vision in Children
Keywords: biofeedback; vision rehabilitation; nystagmus; paediatric
MeSH Terms: conditions — Nystagmus, Pathologic

STUDY DESIGN:
Intervention Model Description: A prospective randomized controlled parallel group study ratio 1:1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (treatment) (Active Comparator): Each session includes 20 minutes of training each with rest as needed. The procedure involves presentation of a standard LED fixation target (FT) consisting of a small red circle of about 0.76° diameter. A fixation training target (FTT) will be selected by the trainer at a perceived better fixation point. Initially the participant will be instructed to stare at the FT circle. Following this stage the participant will be guided to look in the direction of the FTT and listen simultaneously to the audio feedback. As performing this task, the participant will actively control the eye movements until the audio feedback becomes more frequent and then becomes a continuous sound pattern. This continuous sound will signalize to the patient that the FTT location was reached. Participants will be given take-home efficiency reading exercises.
  Interventions: Device: Biofeedback Training
- Group B (control) (Sham Comparator): The simulated biofeedback training for Group B involves the following procedure:
  For four weeks, presentation of a C10-2 microperimetry program. The procedure involves presentation of a standard LED fixation target (FT) consisting of a small red circle of about 0.76° diameter. Initially the participant will be instructed to stare at the FT circle. Following this stage the participant will be guided to look at the FT and simultaneously to be aware of any flashing lights in the periphery of vision. As performing this task, the participant will actively control the eye movements and similar to computer games, the patient has to identify targets in the peripheral field of vision and respond by pressing a button. Participants will be given take-home efficiency reading exercises.
  Interventions: Device: Sham - simulated BT

INTERVENTIONS:
Device: Biofeedback Training — Microperimeter biofeedback training as described provides to the patient a variable frequency sound and a luminous stimulus that vary according to the eyes position, thus guides the oculomotor control and fixation stability accordingly.
  Arms: Group A (treatment)
Device: Sham - simulated BT — The simulated biofeedback training for Group B involves the following: each session includes presentation of a C10-2 microperimetry program. The procedure involves presentation of a standard LED fixation target (FT) consisting of a small red circle of about 0.76° diameter. Initially the participant will be instructed to stare at the FT circle. Following this stage the participant will be guided to look at the FT and simultaneously to be aware of any flashing lights in the periphery of vision. As performing this task, the participant will actively control the eye movements and similar to computer games, the patient has to identify targets in the peripheral field of vision and respond by pressing a button.
  Arms: Group B (control)

SUMMARY:
Active eye movement control training, an old and still most prevalent intervention in low vision rehabilitation (LVR) was never used in nystagmus clinically.

Biofeedback training (BT) is the latest and newest technique for oculomotor control training in cases with low vision when using available modules in the new microperimetry instruments. Laboratory studies in the literature highlighted positive benefits from using BT in nystagmus cases. The purpose of this study is to assess systematically the impact of BT in a series of cases with Infantile Idiopathic Nystagmus (IIN) and formulate guidelines for further use of this intervention in nystagmus cases in general.

DETAILED DESCRIPTION:
Background:

Infantile idiopathic nystagmus (IIN) or congenital motor nystagmus is most common among infantile nystagmus cases. It has a characteristic waveform eye movement pattern with an exponentially increasing velocity slow-phase followed by a saccadic fast phase.

IIN is present from infancy but usually recognized few months into life and may even be evident only after the child has reached several years of age. Characteristics of IIN include the following: conjugate eye movements with equal frequency and amplitude in each eye, gaze position does not change the direction of fast phase, a null point may be present with less motor instability, convergence achieves better motor stability, head turn and head tilt present to facilitate viewing at null point and absence of oscillopsia in most cases.

When the patient is asymptomatic no treatment is required. However, if the visual acuity is decreased with abnormal head posture and oscillopsia interventions are warranted.

Traditional used therapies include muscle surgery, optical devices, drugs and botulinum toxin injections. All current available therapies aim at changing the functional balance among eye muscles responsible for eye movements with hope that they will produce better ocular stability and better foveation time for incoming images with better vision. All such cases also require Low Vision Rehabilitation interventions to improve functional vision and Quality of Life.

Rationale for the study:

Active eye movement control training, an old and still most prevalent intervention in low vision rehabilitation (LVR) was never used in nystagmus cases with low vision for various reasons. One of them was the inability to document accurately eye movements and fixation characteristics in patients with low vision, nystagmus cases included.

Biofeedback training (BT) is the latest and newest technique for oculomotor control training in cases with low vision when using available modules in the new microperimetry instruments.

Sporadic reports in the literature highlighted positive benefits from using BT in a variety of nystagmus cases. The purpose of this study is to assess systematically the impact of BT in a series of cases with IIN and formulate guidelines for further use of this intervention in nystagmus cases in general.

Study hypothesis

The visual and audio parts of the BT program improve in a synergistic way oculomotor control through attention improvement and volitional eye movements towards pre-designated targets. Improved oculomotor control results in better fixation stability of eyes. Better fixation stability in turn results in better vision for distance and near. Dual sensory BT is a therapy used in low vision for more than ten years, showing good results for near and distance vision in cases with macular degeneration and other pathologies. The study hypothesis, never tested before, is that BT in cases with IIN will impact positively oculomotor control and visual acuity as it was proven to do in cases with macular degeneration.

Significance of the study:

Most cases with IIN suffer also from poor visual acuity and in essence are visually impaired. Where as in cases with visual impairment near vision can be easily improved to functional levels using magnification in spectacle glasses, distance vision cannot be improved further with spectacle glasses and other low vision devices are required. BT in IIN cases may result in significant improvement in visual abilities for distance in a similar way that BT results in improved distance vision in cases with macular degeneration.

Clinical trial design:

This is prospective clinical randomized trial to include a control group and take place over a period of up to 24 months.

The objectives set for this trial is to verify if BT impacts on oculomotor control in cases with IIN and results in better distance visual acuity in those trained with BT.

Clinical trial population:

The intended population for this clinical trial is to be found among the Low Vision Rehabilitation (LVR) clinical practice patients. Patients will be considered for inclusion into the study if they meet the trial entry criteria.

The following is an overview of the study procedures: following obtaining consent from study participants, confirmation of eligibility, and baseline assessments (Visit1, V1), participants will undergo 4 BT sessions (V2, V3, V4 and V5). Upon completion of the 4 BT sessions participants will return for a follow up after 1 week (V6) and 3 months (V7).

Baseline procedures During the baseline visit (Visit 1) participants will be assessed for Best Corrected Visual Acuity (BCVA) for distance vision with ETDRS charts at 4 meters, preferred retinal locus (PRL) characteristics, fixation stability (FS) estimates and nystagmus amplitude with the MAIA microperimeter (Centervue, Padova, Italy). Participants will be assessed also for near vision and contrast sensitivity measured with the 2 contrast levels Colenbrander chart, stereopsis will be assessed with the Frisby Stereo Test and Quality of Life estimates will be assessed with the children's visual function questionnaire (CVFQ).

This visit may take an hour time. Training procedure during training procedure visits (V2-5) the participant is seated in front of the instrument while visual targets are presented to the eye and auditory stimuli are presented in tandem with the visual stimuli. Patient has to identify targets and respond by pressing a button.

BT includes 4 BT attempts of 5 minutes each with 5 minutes rest time between each attempt. The procedure involves presentation of a standard LED fixation target (FT) consisting of a small red circle of about 0.76° diameter. A fixation training target (FTT) will be selected by the trainer at a perceived better fixation point. Initially the participant will be instructed to stare at the FT circle. Following this stage, the participant will be guided to look in the direction of the FTT and listen simultaneously to the audio feedback. As performing this task, the participant will actively control the eye movements until the audio feedback becomes more frequent and then becomes a continuous sound pattern. This continuous sound will signalize to the patient is controlling nystagmus.

Simulated BT includes presentation of a C10-2 microperimetry program. The procedure involves presentation of a standard LED fixation target (FT) consisting of a small red circle of about 0.76° diameter. Initially the participant will be instructed to stare at the FT circle. Following this stage, the participant will be guided to look at the FT and simultaneously to be aware of any flashing lights in the periphery of vision. As performing this task, the participant will actively control the eye movements and similar to computer games, the patient has to identify targets in the peripheral field of vision and respond by pressing a button.

Participants will be given take-home efficiency reading exercises. Training visits are repeated to a total of 4 on a weekly interval.

End of study procedures Additional follow up Visits 6 and 7 will take place at 5 weeks and 4 months following visit 1. Participants will be assessed also for near vision and contrast sensitivity measured with the 2 contrast levels Colenbrander chart, stereopsis will be assessed with the Frisby Stereo Test and Quality of Life estimates will be assessed with the children's visual function questionnaire (CVFQ).

There are no known risks or side effects known from using biofeedback training. In some cases, perceived side effects observed are general fatigue, tiredness due to the efforts to fixate, discomfort or eye strain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as Infantile idiopathic nystagmus (IIN)
* Ability to follow the visual and auditory stimuli and training instructions

Exclusion Criteria:

* Ocular diseases not related to the nystagmus physiopathology
* Both eyes with media opacity that impairs microperimetry testing
* Peripheral nystagmus cases
* Other types of nystagmus than IIN
* Inability to perform during testing and training

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Best Corrected Visual Acuity for Distance Vision across BT sessions and post BT | 7 days from baseline (V2), 14 days (V3), 21 days (V4), 28 days (V5), 35 days (V6), and 118 days from baseline (V7)
  Measured with the ETDRS charts at 4 m
Changes in Fixation Stability (Bivariate contour ellipse area) across BT sessions and post BT | 7 days from baseline (V2), 14 days (V3), 21 days (V4), 28 days (V5), 35 days (V6), and 118 days from baseline (V7)
  Represents the area used for fixation on the retina in square degrees as given by the microperimeter

SECONDARY OUTCOMES:
Changes in Contrast Sensitivity for near vision across BT sessions and post BT | 35 days from baseline (V6), and 118 days from baseline (V7)
  Two contrast Colenbrander chart
Changes in Stereopsis for near vision across BT and post BT | 35 days from baseline (V6), and 118 days from baseline (V7)
  Frisby Stereotest for near with best near correction
Changes in Quality of Life Parental Questionnaire across BT and post BT | 35 days from baseline (V6), and 118 days from baseline (V7)
  Quality of Life estimates will be assessed with the children's visual function questionnaire (CVFQ).(16)
Changes in Reading speed across BT sessions and post BT | 35 days from baseline (V6), and 118 days from baseline (V7)
  Using the MNRead Test with the best near correction

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Markowitz, MD, Principal Investigator — University of Toronto
Locations (1):
- CNIB, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abadi RV, Bjerre A. Motor and sensory characteristics of infantile nystagmus. Br J Ophthalmol. 2002 Oct;86(10):1152-60. doi: 10.1136/bjo.86.10.1152. PMID 12234898
- [Background] Rucker JC. Current Treatment of Nystagmus. Curr Treat Options Neurol. 2005 Jan;7(1):69-77. doi: 10.1007/s11940-005-0008-0. PMID 15610709
- [Background] ANDERSON JR. Causes and treatment of congenital eccentric nystagmus. Br J Ophthalmol. 1953 May;37(5):267-81. doi: 10.1136/bjo.37.5.267. No abstract available. PMID 13042022
- [Background] KESTENBAUM A. [New operation for nystagmus]. Bull Soc Ophtalmol Fr. 1953 Jun;6:599-602. No abstract available. Undetermined Language. PMID 13115959
- [Background] Wang ZI MS, Dell'Osso LF , Ph.D. A Review of the Tenotomy Nystagmus Surgery: Origin, Mechanism, and General Efficacy. Neuro-Ophthalmology, 31:157-165, 2007 ISSN: 0165-8107 DOI: 10.1080/01658100701647704
- [Background] Yaniglos SS, Stahl JS, Leigh RJ. Evaluation of current optical methods for treating the visual consequences of nystagmus. Ann N Y Acad Sci. 2002 Apr;956:598-600. doi: 10.1111/j.1749-6632.2002.tb02893.x. No abstract available. PMID 11960878
- [Background] Lennerstrand G, Nordbo OA, Tian S, Eriksson-Derouet B, Ali T. Treatment of strabismus and nystagmus with botulinum toxin type A. An evaluation of effects and complications. Acta Ophthalmol Scand. 1998 Feb;76(1):27-7. doi: 10.1034/j.1600-0420.1998.760106.x. PMID 9541431
- [Background] Buia C, Tiesinga P. Attentional modulation of firing rate and synchrony in a model cortical network. J Comput Neurosci. 2006 Jun;20(3):247-64. doi: 10.1007/s10827-006-6358-0. Epub 2006 Apr 22. PMID 16683206
- [Background] Shtark MB, Kozlova LI, Bezmaternykh DD, Mel'nikov MY, Savelov AA, Sokhadze EM. Neuroimaging Study of Alpha and Beta EEG Biofeedback Effects on Neural Networks. Appl Psychophysiol Biofeedback. 2018 Jun;43(2):169-178. doi: 10.1007/s10484-018-9396-2. PMID 29926265
- [Background] Markowitz SN, Reyes SV. Microperimetry and clinical practice: an evidence-based review. Can J Ophthalmol. 2013 Oct;48(5):350-7. doi: 10.1016/j.jcjo.2012.03.004. Epub 2012 Oct 23. PMID 24093179
- [Background] Nido MD, Markowitz SN. Vision rehabilitation with biofeedback training. Can J Ophthalmol. 2018 Jun;53(3):e83-e84. doi: 10.1016/j.jcjo.2017.11.003. Epub 2017 Dec 21. No abstract available. PMID 29784180
- [Background] Ciuffreda KJ, Goldrich SG, Neary C. Use of eye movement auditory biofeedback in the control of nystagmus. Am J Optom Physiol Opt. 1982 May;59(5):396-409. doi: 10.1097/00006324-198205000-00007. PMID 7102798
- [Background] Grenga PL, Trabucco P, Meduri A, Fragiotta S, Vingolo EM. Microperimetric biofeedback in a patient with oculocutaneous albinism. Can J Ophthalmol. 2013 Oct;48(5):e105-7. doi: 10.1016/j.jcjo.2012.11.011. Epub 2013 Aug 29. No abstract available. PMID 24093197
- [Background] Mezawa M, Ishikawa S, Ukai K. Changes in waveform of congenital nystagmus associated with biofeedback treatment. Br J Ophthalmol. 1990 Aug;74(8):472-6. doi: 10.1136/bjo.74.8.472. PMID 2390522
- [Background] Daibert-Nido M, Patino B, Markowitz M, Markowitz SN. Rehabilitation with biofeedback training in age-related macular degeneration for improving distance vision. Can J Ophthalmol. 2019 Jun;54(3):328-334. doi: 10.1016/j.jcjo.2018.10.016. Epub 2019 Apr 2. PMID 31109472
- [Background] Felius J, Stager DR Sr, Berry PM, Fawcett SL, Stager DR Jr, Salomao SR, Berezovsky A, Birch EE. Development of an instrument to assess vision-related quality of life in young children. Am J Ophthalmol. 2004 Sep;138(3):362-72. doi: 10.1016/j.ajo.2004.05.010. PMID 15364217